CLINICAL TRIAL: NCT01151787
Title: Efficacy and Safety of Cyclobenzaprine Hydrochloride Extended Release for the Treatment of Chronic Migraine: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Efficacy and Safety of Cyclobenzaprine Hydrochloride Extended Release for the Treatment of Chronic Migraine
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was never initiated under new location/provider group. Contract to continue was never signed between TEVA and Kennedy Headache Center
Sponsor: Kennedy Medical Group (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CEPH03242010
Record Dates: First submitted 2010-06-25; First posted 2010-06-28 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Migraine
Keywords: migraine
MeSH Terms: conditions — Migraine Disorders | interventions — cyclobenzaprine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cyclobenzaprine hydrochloride (Active Comparator)
  Interventions: Drug: cyclobenzaprine hydrochloride
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: cyclobenzaprine hydrochloride — 15mg daily for 3 months
  Other Names: cyclobenzaprine hydrochloride is Amrix 15mg/daily
  Arms: cyclobenzaprine hydrochloride
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
The primary objective of the study is to evaluate the effectiveness and safety of cyclobenzaprine hydrochloride extended release (Amrix 15mg/day) for the prophylaxis of chronic migraine compared to a placebo medication. A second objective, is to find out whether there is an improvement in quality of sleep and self-reported depression in patients taking Amrix 15mg daily. The hypothesis is that the number of migraine days per month of patients treated with Amrix 15mg daily will be significantly lower than those patients treated with placebo.

ELIGIBILITY:
Inclusion Criteria:

1. males and females, aged 18 to 65, with headaches longer than 30 minutes per day for at least 15 days per month (28 days) meeting ICHD-IIR criteria for chronic migraine. Subjects must have headaches at least 8 days per month which are alleviated with triptans or ergots AND/OR which have at least 1 migrainous feature (unilaterality of headache or pain more prominent on 1 side of the head, throbbing, nausea, vomiting, photophobia, phonophobia, increased pain with physical exertion or avoidance of exertion)
2. subjects willing and able to perform all study-related measures including accurately completing study diaries and instruments, maintaining stable doses of headache preventative medications, completing study visits and obtaining blood testing as indicated.
3. women of childbearing potential must use an acceptable method of birth control for the duration of the study (oral contraceptives, IUD, injectable or intravaginal contraception or barrier methods combined with spermicide)

Exclusion Criteria:

1. subjects <18 and >65 years of age
2. pregnancy or attempted pregnancy during the study
3. nursing females
4. psychiatric condition which, in the investigator's opinion will influence trial safety or data collection
5. new daily persistent headache, hemicrania continua, chronic tension-type headache or cluster headache diagnoses.
6. headache suspicious for and not investigated to rule out secondary headache disorder
7. angle closure glaucoma
8. urinary retention
9. hepatic impairment felt by the investigator to interfere with study safety (as determined from history and/or prerequisite liver function testing within 1 year of study enrollment)
10. within 14 days of MAO inhibitor use or discontinuation
11. known hypersensitivity to cyclobenzaprine hydrochloride or any component of Amrix formulation
12. concomitant tramadol or tricyclic antidepressant use
13. history of myocardial infarction or congestive heart failure
14. hyperthyroidism
15. new start of daily preventative medication (which may influence headaches) less than 2 months preceding enrollment
16. dosage change or discontinuation of daily preventative medication (which may influence headaches) within 1 month of trial enrollment -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Mean total number of migraine/migrainous headache days per month | 4 months
  The principle outcome variable will be the mean total number of migraine/migrainous headache days which will be calculated for the month prior to enrollment in the study (pretreatment) and then calculated for the third month after study treatment (posttest) after taking 15mg of Amrix or the placebo.

SECONDARY OUTCOMES:
Mean total number of headache days/month | 4 months
mean peak daily and mean average daily pain intensity ratings/month | 4 months
mean total number of abortive treatment days/month | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Loretta Mueller, DO, Principal Investigator — Kennedy Medical Group dba The Headache Center at Kennedy Health Alliance
Locations (1):
- The Headache Center at Kennedy Health Alliance, Cherry Hill, New Jersey, United States